CLINICAL TRIAL: NCT01904994
Title: LINK4HEALTH: A Combination Approach to Linkage and Retention for HIV (Human Immunodeficiency Virus) Infected Individuals in Swaziland
Brief Title: Link4Health: A Combination Strategy for Linkage and Retention, Swaziland
Acronym: L4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAL2708; 5R01AI100059-02 (NIH)
Record Dates: First submitted 2013-07-16; First posted 2013-07-22 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: HIV (Human Immunodeficiency Virus); ART (antiretroviral therapy); financial incentive; linkage; retention; SMS (Short Message Service) appointment reminder; accelerated ART; CD4+ count
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Point-of-Care Systems; Potassium Iodide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Participants will be managed per standard of care following prevailing Swaziland Ministry of Health guidelines.
- Combined Intervention Strategy (Experimental): Point-of-care (POC) CD4+ (cluster of differentiation 4) Count Accelerated ART initiation for ART eligible participants Basic care and prevention package Cellular Appointment Reminders and Follow-Up Financial Incentives
  Interventions: Procedure: POC (point-of-care) CD4+ (cluster of differentiation 4) Count; Procedure: Accelerated ART (antiretroviral therapy) Initiation; Behavioral: Basic Care and Prevention Package; Behavioral: Cellular Appointment Reminders and Follow-Up; Other: Financial Incentive

INTERVENTIONS:
Procedure: POC (point-of-care) CD4+ (cluster of differentiation 4) Count — Each HIV testing and counseling (HTC) site will be equipped with POC CD4+ testing using PIMA™ Analyser (Inverness), test strips, and reagents. Study staff will obtain 25 microliters of blood via finger prick and process the POC (point-of-care) CD4+ (cluster of differentiation 4) Count' test immediately following the baseline interview. Test results will be recorded on study forms including a referral form that has multiple copies, one copy to be given to the participant, the second sent to the affiliated HIV (Human immunodeficiency virus)care clinic in the study unit, and the third kept by study staff in a locked cabinet with other confidential material. All participants, regardless of the CD4+ result, will be encouraged to enroll in HIV care as soon as they can.
  Other Names: PIMA
  Arms: Combined Intervention Strategy
Procedure: Accelerated ART (antiretroviral therapy) Initiation — Accelerated ART initiation for patients with POC CD4+ < 350 cells/uL (micro-liter) within 1 week from testing.
  2 counseling sessions (one at time of HTC and other at first HIV clinic visit), and collection of blood for other baseline lab tests, but initiation prior to return of results for patients who do not meet criteria for waiting
  Arms: Combined Intervention Strategy
Behavioral: Basic Care and Prevention Package — Basic care and prevention package (BCPP) provided approximately every three months that includes: condoms; soap, pill box and pictorial education about use of materials and HIV, such as family testing tools and information. Information on BCPP contents and review the educational materials will be provided. An example of educational materials is a family-testing tool to encourage the participant to have all family members tested for HIV. All BCPP items will be replenished every 3 months for all participants, regardless of ART status, beginning at linkage to HIV care.
  Other Names: BCPP
  Arms: Combined Intervention Strategy
Behavioral: Cellular Appointment Reminders and Follow-Up — SMS (short messaging service) appointment reminders for follow-up appointments.
  Telephone call within 7 days of missed appointment for all patients.
  Arms: Combined Intervention Strategy
Other: Financial Incentive — Participants will receive a series of financial incentives to support linkage into care within 1 month and retention in care at 6 months and 12 months after testing HIV positive. The value of the financial incentive (FI) will be 80 Swaziland Rand, calculated based on the associated financial costs of traveling to clinic. These incentives will be distributed by through mobile airtime. Participants without mobile phones will be given an alternative incentive of equal value, such as a store voucher.
  Other Names: FI (Financial Incentive)
  Arms: Combined Intervention Strategy

SUMMARY:
Despite increased HIV (Human Immunodeficiency Virus) infection testing in Africa, many patients never enroll in subsequent HIV care after testing or remain in care after an initial enrollment. This study's aim is to improve linkage to HIV care and retention in HIV care through the use of feasible, evidence-based, and practical interventions. The study takes place in Swaziland, the country with the highest HIV prevalence (24%) in sub-Saharan Africa. The study will randomize groups of HIV testing sites and affiliated clinics to either standard of care or a combined intervention strategy (CIS) which consists of point-of care CD4 (cluster differentiation 4 (CD4)) testing at time of HIV testing, fast-track HIV medications for those who are eligible for treatment,mobile phone appointment reminders, care bags filled with health prevention materials, and financial incentives. The study outcomes are linkage to and retention in care as well as cost effectiveness, feasibility of interventions, and patient acceptability of interventions.

DETAILED DESCRIPTION:
Linkage of patients from HIV testing to HIV care programs and their retention once enrolled in care are essential to HIV program effectiveness in terms of prevention of HIV;related morbidity and mortality and prevention of HIV transmission. Linkage and retention rates in HIV programs in sub-Saharan Africa (SSA) are suboptimal, with less than half of patients who test positive successfully linking and remaining in care at 1 year. This study is a two-arm cluster site;randomized trial to compare the effectiveness of a novel combination package of evidence;based interventions, the combination intervention strategy (CIS), compared to standard of care (SOC) on linkage and retention of HIV;positive patients from point of testing to retention in care. CIS will include 1) point of care CD4+ count assays at HIV testing sites; 2) accelerated antiretroviral therapy (ART) initiation for eligible patients; 3) provision of a basic care and prevention package (BCPP); 4) short message service (SMS) reminders for clinic appointments; and 5) financial incentives for linkage and retention. The primary aim is to evaluate the effectiveness of CIS as compared to SOC on the combined outcome of rapid linkage to HIV care within 1 month and retention in care at 12 months among adults testing positive for HIV. Secondary aims include evaluation of the effectiveness of CIS compared to SOC on each of linkage to HIV; retention in care; time to ART initiation; HIV disease progression and mortality; patient acceptability; association between baseline characteristics and outcomes, and comparison of cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Testing HIV-positive at an HTC (HIV testing and counseling) site within a SU (study unit)
* Willing to be referred to an HIV care clinic associated with the SU
* Willing to provide locator information
* Willing to adhere to study procedures, including a baseline interview, home-based interviews at 1 and 12 months after study enrollment; home-based CD4+ count assessment 12 months after enrollment, and abstraction of data from their medical records.
* Able to provide informed consent

Exclusion Criteria:

* Planning on leaving the community where they currently reside in the next 12 months for a period greater than 6 months
* Enrolled in HIV (Human immunodeficiency virus) care in the past 6 months at any HIV care clinic
* Currently on ART (antiretroviral therapy)
* Initiated ART (for any duration) in the past 6 months at any HIV care clinic
* Does not speak or understand English or si-Swati
* Reports being currently pregnant at time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2201 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Change in proportion of participants who both link to care at assigned study unit within 1 month and are retained in care at the designated study unit 12 months after HIV (Human Immunodeficiency Virus) diagnosis | one month after enrollment, 12 months after enrollment
  Combined outcome of linkage to HIV care within 1 month after testing HIV positive and retention in care 12 months after testing.
  Participants are considered to achieve this outcome if they successfully link to the HIV clinic at their study unit (SU) within 1 month of testing HIV positive and are retained in care at the HIV clinic at their SU 12 months after testing HIV positive, as measured from medical records.

SECONDARY OUTCOMES:
Proportion of participants successfully linked to care at designated study unit within 1 month of HIV diagnosis | 12 months after enrollment
  Linkage to care within 1 month of HIV testing (at any clinic within the assigned study unit).
Proportion of participants retained in care at designated study unit 12 months after HIV diagnosis. | 12 months after enrollment
  Retention in care 12 months after HIV testing, independent of linkage at 1 month (at any clinic within the assigned study unit).
Change in proportion of participants successfully linked to care at any HIV care clinic within one month of HIV diagnosis | one month after enrollment, 12 months after enrollment
  Proportion of participants successfully linked to care at any HIV care clinic within one month of HIV diagnosis
Median time from HIV testing to initial assessment of ART (antiretroviral) eligibility | 12-months after enrollment
  Time from linkage to ART eligibility assessment
Median time from HIV testing to ART eligibility | 12 months after enrollment
  Time from HIV testing to ART eligibility
Proportion of participants who consistently engage in care (attend > 75% of scheduled appointments) | 12-months after enrollment
  Proportion of participants who consistently engage in care, defined as attend > 75% of scheduled appointments
Change in proportion of participants with new World Health Organization (WHO) Stage III/IV event or hospitalization | 1 month after enrollment,12 months after enrollment
  Proportion of participants with new WHO Stage III/IV event or hospitalization
Median CD4+ (cluster difference 4) count and viral load 12 months after HIV diagnosis | 12 months after testing HIV-positive
  Median CD4+ cell count 12 months after HIV diagnosis, median viral load 12 months after HIV diagnosis
Change in Mortality rate | 1 month after enrollment, 12 months after enrollment
  Mortality rate 12 months after HIV diagnosis
Change in proportion of participants reporting interventions were received | 1 month after enrollment, 12 months after enrollment
  Proportion of participants, who are randomized to study units receiving CIS, reporting receipt of each intervention
Proportion of participants reporting that interventions were highly acceptable | 12 months after enrollment
  Proportion of participants, who are randomized to study units receiving CIS, reporting that interventions were highly acceptable

OTHER OUTCOMES:
Change in adjusted risk ratio comparing proportion of participants who both link to care at assigned study unit within one month and are retained in care at designated study unit twelve months after HIV diagnosis | at enrollment, one month after enrollment, 12 months after enrollment
  Adjusted risk ratio comparing proportion of participants who both link to care at assigned study unit within one month and are retained in care at designated study unit twelve months after HIV diagnosis, by strata of age, sex, and other socio-demographic variables

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa El-Sadr, MD MPH, Principal Investigator — ICAP Columbia University; Charles Azih, MD MPH, Study Director — Swaziland MOH; Scott Braithwaite, MD MSc, Study Director — New York University; Batya Elul, PhD MD, Study Director — ICAP Columbia University; Peter Ehrenkranz, MD MPH, Study Director — Centers for Disease Control and Prevention; Matthew Lamb, PhD MPH, Study Director — ICAP Columbia University; Margaret McNairy, MD MSc, Study Director — ICAP Columbia University; Phumzile Mndzebele, Study Director — Swaziland MOH; Ruben Sahabao, MD, Study Director — ICAP Swaziland
Locations (20):
- Eswatini (20):
  - Bhalekane Clinic, Swaziland
  - Dvokolwako, Swaziland
  - Good Shepherd Hospital, Swaziland
  - Hlatikhulu Hospital, Swaziland
  - Horo, Swaziland
  - Kamfishane, Swaziland
  - Lamvelase, Swaziland
  - Luyengo Clinic, Swaziland
  - Mangweni Clinic, Swaziland
  - Mankayane Hospital, Swaziland
  - Mashobneni Clinic, Swaziland
  - Mbabane Government Hospital, Swaziland
  - Mkhuzweni Health Center, Swaziland
  - Motshane, Swaziland
  - Mpolenjeni Clinic, Swaziland
  - Nhlangano Health Center, Swaziland
  - Piggs Peak, Swaziland
  - Raleigh Fitkin Memorial Hospital, Swaziland
  - Siphofaneni Clinc, Swaziland
  - Sithobeloa Rural Health Center, Swaziland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McNairy ML, Lamb MR, Gachuhi AB, Nuwagaba-Biribonwoha H, Burke S, Mazibuko S, Okello V, Ehrenkranz P, Sahabo R, El-Sadr WM. Effectiveness of a combination strategy for linkage and retention in adult HIV care in Swaziland: The Link4Health cluster randomized trial. PLoS Med. 2017 Nov 7;14(11):e1002420. doi: 10.1371/journal.pmed.1002420. eCollection 2017 Nov. PMID 29112963
- [Derived] McNairy ML, Gachuhi AB, Lamb MR, Nuwagaba-Biribonwoha H, Burke S, Ehrenkranz P, Mazibuko S, Sahabo R, Philip NM, Okello V, El-Sadr WM. The Link4Health study to evaluate the effectiveness of a combination intervention strategy for linkage to and retention in HIV care in Swaziland: protocol for a cluster randomized trial. Implement Sci. 2015 Jul 19;10:101. doi: 10.1186/s13012-015-0291-4. PMID 26189154